CLINICAL TRIAL: NCT06970392
Title: Brief Sleep Intervention for Bedtime Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Andrew Riley, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00025469
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Child Sleep
Keywords: Feasibility trial; Bedtime Resistance; Bedtime Pass; Primary Care; Integrated Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bedtime Pass (Experimental): The behavioral health consultant will converse with the participant about the child's bedtime resistance, bedtime routine, and other variables that may impact sleep. The behavioral health consultant will provide psychoeducation on sleep hygiene and provide relevant handouts. The behavioral health consultant will also explain the Bedtime Pass Intervention and provide relevant materials. The participant will have the opportunity to ask questions about implementing the intervention at home with their child.
  Interventions: Behavioral: Bedtime Pass

INTERVENTIONS:
Behavioral: Bedtime Pass — The Bedtime Pass is a small paper card that children will be allowed to exchange for a trip out of their bedroom after bedtime. Once the card has been exchanged, participants will be instructed to ignore any additional pleas from their child. Participants will also be provided with general information about good sleep hygiene.

SUMMARY:
This is non-controlled feasibility study testing the delivery of a brief sleep intervention for children aged 3-7 who struggle to fall asleep independently. The interventions is designed to be delivered by a behavioral health consultant during routine primary care visits. The treatment components consist of education about good sleep hygiene and the "Bedtime Pass." The hypotheses are that the intervention will be delivered with fidelity in the time allotted, and that parents will rate the intervention as feasible and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a child aged 3-7 years who receives primary care services who endorses their child demonstrating bedtime resistance; English-speaking; receiving primary care at the study locations.

Exclusion Criteria:

* Existing receipt of more intensive sleep intervention; severe intellectual disability or other condition precluding participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability Survey | Immediately post-intervention and 30 days post-intervention
Treatment Fidelity Checklist | Immediately post-intervention

SECONDARY OUTCOMES:
Pediatric Insomnia Severity Index | 30 days post-intervention

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be available from the PI upon request .
Supporting Information: Study Protocol
Time Frame: 5 years from the end of the study.
Access Criteria: Anonymized data will be available from the PI upon request.